CLINICAL TRIAL: NCT05391750
Title: A Phase 1 Study Evaluating the Safety of Venetoclax and Tocilizumab in African American and Non-African American Subjects With Relapsed or Refractory t(11;14) Multiple Myeloma
Brief Title: Venetoclax and Tocilizumab for the Treatment of Patients With Relapsed or Refractory t(11;14) Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathan Kaufman, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002448; NCI-2021-02510 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002448; WINSHIP5273-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-05-26 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab; Immunoglobulin G; Disulfides; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, tocilizumab) (Experimental): Patients receive tocilizumab IV on day -7 of cycle 1, and on day 1 of subsequent cycles. Patients also receive venetoclax PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Tocilizumab; Drug: Venetoclax

INTERVENTIONS:
Biological: Tocilizumab — Given IV
  Other Names: Actemra; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA; R-1569; RoActemra
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial finds out the best dose and side effects of venetoclax and tocilizumab in treating patients with t(11;14) multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Tocilizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Tocilizumab is used to treat side effects from immune therapy in patients with myeloma. Giving venetoclax and tocilizumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the dose limiting toxicity (DLT), safety profile, and the recommended phase 2 dose (RPTD) of venetoclax and tocilizumab when administered in subjects with relapsed and recurrent (RR) multiple myeloma t(11;14) (MM).

SECONDARY OBJECTIVES:

I.To evaluate the preliminary efficacy data regarding the effect of venetoclax and tocilizumab by objective response rate per IMWG criteria.

II. To evaluate the effect of chronic tocilizumab administration on venetoclax exposure.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To evaluate the preliminary efficacy data regarding the effect of venetoclax and tocilizumab by time to response (TTR), time to disease progression (TTP), duration of response (DOR), progression free survival (PFS) and overall survival (OS).

II. To measure the effect of IL6 receptor blockade on ex vivo venetoclax sensitivity.

III. To evaluate the cell populations in the bone marrow of responders versus non-responders as well as the effect of IL6 receptor blockade on those populations.

IV. To evaluate the expression of B cell markers on venetoclax sensitive myeloma.

V. To determine the expression of key BCL2 family members with and without IL6 receptor blockade.

VI. To correlate differences in somatic mutations, structural alterations, gene expression and chromatin accessibility with venetoclax response.

OUTLINE: This is a dose-escalation study of venetoclax and tocilizumab.

Patients receive tocilizumab intravenously (IV) on day -7 of cycle 1, and on day 1 of subsequent cycles. Patients also receive venetoclax orally (PO) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks, then every 6 months thereafter.

ELIGIBILITY:
Subject must be >= 18 years of age Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of =< 2

Diagnosis of multiple myeloma that requires treatment and has been previously treated with:

* Has received at least 2 prior lines of therapy
* Has had documented disease progression on or within 60 days after completion of the last therapy.
* Has received at least 2 consecutive cycles of lenalidomide and be relapsed/refractory to lenalidomide, as defined per protocol.
* Has received at least 2 consecutive cycles of a proteasome inhibitor (PI). Have MM positive for t(11;14) translocation as determined by an analytically validated fluorescence in-situ hybridization (FISH) assay per the central laboratory testing

Subject must have had measurable disease at Screening, defined as any of the following:

* Serum monoclonal protein >= 1.0 g/dL (>= 10 g/L) by protein electrophoresis, or
* >= 200 mg of monoclonal protein in the urine on 24-hour electrophoresis, or
* Serum immunoglobulin free light chain (FLC) >= 10 mg/dL provided serum FLC ratio is abnormal

Subjects with a history of autologous transplantation must have adequate peripheral blood counts as defined below, have recovered from any transplant related toxicity(s) and be > 100 days post-autologous transplant (prior to first dose of study drug)

Subjects must meet the following laboratory parameters, per laboratory reference range, at least once during the screening period:

* Absolute neutrophil count (ANC) >= 1000/uL (Subject may use granulocyte colony-stimulating factor [G-CSF] to achieve ANC eligibility criteria)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x upper limit of normal range (ULN)
* Calculated creatinine clearance >= 30 mL/min using a modified Cockcroft- Gault calculation or a 24-hour urine collection for creatinine clearance
* Platelet count >= 75,000 cells/mm3 and independent of transfusion for 2 weeks
* Hemoglobin >= 8.0 g/dL, subjects may not receive blood transfusion within 1 week to achieve hemoglobin eligibility criteria per investigator discretion
* Total bilirubin =< 1.5 x ULN; subjects with Gilbert's syndrome may have bilirubin > 1.5 x ULN

If female, subject must be:

* Postmenopausal defined as:

  * Age > 55 years with no menses for 24 or more months without an alternative medical cause
  * Age =< 55 years with no menses for 24 or more months without an alternative medical cause
  * AND an follicle stimulating hormone (FSH) level > 40 IU/L. OR
* Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) OR
* A woman of childbearing potential (WOCP) practicing at least one protocol specified method of birth control starting at cycle 1 day 1 (or earlier) through at least 30 days after last dose of study drug

  * Females of childbearing potential (must have negative results for pregnancy test performed:
* At screening, on a serum or urine sample obtained within 28 days prior to the first study drug administration,
* Prior to dosing, on a urine sample obtained on the first day of study drug dosing, if it has been > 7 days since obtaining the serum pregnancy test results
* Females of non-childbearing potential (either postmenopausal or permanently surgically sterile as defined above) at screening do not require pregnancy testing

Must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

Subject exhibits evidence of other clinically significant uncontrolled condition(s), including, but not limited to:

* Acute infection within 14 days prior to first dose of study drug requiring antibiotic, antifungal, or antiviral therapy
* Diagnosis of fever and neutropenia within 1 week prior to first dose of study drug

Subject has a cardiovascular disability status of New York Heart Association class >= 3

Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular or hepatic disease within the last 6 months that, in the opinion of the investigator, would adversely affect his/her participation in the study

Subject has a history of other active malignancies other than multiple myeloma within the past 3 years prior to study entry, with the following exceptions:

* Adequately treated in situ carcinoma of the cervix uteri,
* Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin,
* Localized prostate cancer Gleason grade 6 or lower AND with stable prostate specific antigen (PSA) levels off treatment
* Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent

Known human immunodeficiency viral (HIV) infection

Active hepatitis B or C infection based on screening blood testing

Subject is receiving other ongoing anti-myeloma therapy

Subject has received any of the following within 7 days prior to the first dose of study drug:

* Strong or moderate CYP3A inhibitors, or
* Strong or moderate CYP3A inducers

Subject has received any of the following within 14 days prior to the first dose of study drug or has not recovered to less than a grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy: any anti-myeloma therapy including chemotherapy, radiotherapy, or investigational therapy, including targeted small molecule agents

Subject has received prior treatment with a BCL-2 family inhibitor

Subject is pregnant, parturient, or breastfeeding; deprived of freedom by judicial or administrative decision; hospitalized and unable to provide consent, or otherwise unable to provide consent

Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit within 3 days prior to the first dose of study drug

Subject has received immunization with live vaccine within 60 days of dosing

Recent corticosteroid therapy at a cumulative dose equivalent to > 140 mg of prednisone or a single dose equivalent to >= 40 mg of dexamethasone within 2 weeks prior to the first dose of study drug

Subject's decision to not divulge the race

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Completion of cycle 1 (each cycle is 21 days)
  The MTD for each arm is selected based on isotonic regression27, using the shiny app BOINComb (http://www.trialdesign.org). The dose is selected as the MTD for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there are ties, the higher dose level is selected when the isotonic estimate is lower than the target toxicity rate; the lower dose level is selected when the isotonic estimate is greater than or equal to the target toxicity rate.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post-treatment
  AEs, related AEs, serious (S)AEs, related SAEs, and AEs leading to interruptions and/or discontinuation of study drug will be analyzed descriptively, using frequencies and percentages.
Overall response rate (ORR) | Up to 5 years
  ORR will be calculated with an exact 95% confidence interval (CI) for each arm, using the Clopper-Pearson method.
Complete response rate | Up to 5 years
  Complete response rate will be calculated with an exact 95% CI for each arm, using the Clopper-Pearson method.
Time to response (TTR) | From date of receipt of study treatment to date of treatment response, where those not responding are censored at date of last follow-up or death from any cause, assessed up to 5 years
  TTR will be estimated using the Kaplan-Meier method. Median TTR will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.
Time to disease progression (TTP) | From date of receipt of study treatment to date of disease progression, where those not progressing or have died are censored at date of last follow-up or death from any cause, assessed up to 5 years
  TTP will be estimated using the Kaplan-Meier method. Median TTP will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.
Duration of response (DOR) | From date of treatment response to date of disease progression, assessed up to 5 years
  Median DOR will be reported, along with the 25th and 75th percentiles.
Progression-free survival (PFS) | From date of receipt of study treatment to date of disease progression or death from any cause, where those alive without are censored at date of last follow-up, assessed up to 5 years
  PFS will be estimated using the Kaplan-Meier method. Median PFS will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.
Overall survival (OS) | From date of receipt of study treatment to date of death from any cause, where those alive without are censored at date of last follow-up, assessed up to 5 years
  OS will be estimated using the Kaplan-Meier method. Median OS will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Kaufman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No